CLINICAL TRIAL: NCT00574600
Title: A Phase 1 Placebo-controlled Clinical Trial to Evaluate the Safety and Immunogenicity of SAAVI DNA-C2 Vaccine Boosted by SAAVI MVA-C Vaccine, in HIV Uninfected Healthy Vaccinia Naive Adult Participants in South Africa and the United States
Brief Title: Safety of and Immune Response to Two HIV Vaccines: SAAVI DNA-C2 Boosted With SAAVIMVA-C, in HIV-Negative Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: HIV Vaccine Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 073/SAAVI 102; 10520 (Registry Identifier: DAIDS ES Registry ID); SAAVI 102; HVTN 073
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccine (Experimental): SAAVI DNA-C2 administered as 1 ml intramuscularly in either deltoid at study entry and Months 1 and 2; SAAVI MVA-C administered as 0.5 ml intramuscularly in either deltoid at Months 4 and 5
  Interventions: Biological: SAAVI DNA-C2 vaccine; Biological: SAAVI MVA-C vaccine
- Placebo (Placebo Comparator): Placebo administered at Months 0, 1, 2, 4 and 5
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: SAAVI DNA-C2 vaccine — DNA vaccine
  Arms: Vaccine
Biological: SAAVI MVA-C vaccine — Boost vaccine
  Arms: Vaccine
Biological: Placebo — Placebo vaccine
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety of and immune response to an experimental DNA HIV vaccine followed by boosting with an experimental modified vaccinia HIV vaccine (MVA) in HIV uninfected adults.

DETAILED DESCRIPTION:
The worldwide HIV/AIDS epidemic may only be controlled through development and utilization of a safe and effective vaccine that will prevent HIV infection. Due to the high prevalence of HIV-1 subtype C in southern Africa, the South African AIDS Vaccine Initiative (SAAVI), the HIV Vaccine Trials Network (HVTN) and the National Institute of Allergy and Infectious Diseases (NIAID) are evaluating two subtype C HIV vaccines, SAAVI DNA-C2 and SAAVI MVA-C through this study . These two vaccines will be used together in a prime-boost regimen. The SAAVI DNA-C2 vaccine is a multigene DNA vaccine consisting of two DNA plasmids in equal amounts that express an HIV-1 subtype C polyprotein comprising of Gag-Reverse Transcriptase-Tat-Nef and an HIV-1 subtype C truncated Env. SAAVI MVA-C is a recombinant MVA vaccine expressing the same immunogens as the SAAVI DNA-C2 vaccine. MVA is a highly attenuated vaccinia virus. The purpose of this study is to evaluate the safety and immunogenicity of an experimental DNA HIV vaccine, SAAVI DNA C2, followed by boosting with an experimental recombinant MVA HIV vaccine, SAAVI MVA-C, in HIV uninfected adults.

Participants will actively participate in this study for 12 months and will then be contacted and asked questions about their health once annually for 3 years following initial study injection. Participants will be randomly assigned to receive either the SAAVI prime-boost preventive vaccine regimen or placebo. Vaccination with the SAAVI DNA-C2 vaccine will occur at Months 0, 1, and 2; boost vaccinations with the SAAVI MVA-C vaccine will occur at Months 4 and 5. Additional study visits will occur at Weeks 2, 6, 10, 16, 18, and 20 and Days 147, 154, 273, and 364.

Study procedures include physical exams, blood and urine collection, HIV testing, an electrocardiogram, and questionnaire. Some blood collected from participants will be stored and used in future research. Risk-reduction counseling will be conducted at all study visits.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory test results within specified ranges [complete blood count, chemistries, cardiac troponin T, urinalysis]
* Good general health
* HIV-1 and -2 uninfected
* Have access to a participating HIV Vaccine Trials Unit (HVTU) and willing to be followed for the duration of the study
* Willing to receive HIV test results
* Negative hepatitis B surface antigen
* Negative hepatitis C virus (HCV) antibodies OR negative HCV PCR if anti-HCV test is positive
* Willing to use acceptable forms of contraception from at least 21 days prior to enrollment through the duration of the study

Exclusion Criteria:

* History of vaccination against smallpox
* HIV vaccines in prior HIV vaccine trial
* Immunosuppressive medications within 168 days prior to first study vaccination
* Blood products within 120 days prior to first study vaccination
* Immunoglobulin within 60 days prior to first study vaccination
* Live attenuated vaccines within 30 days prior to first study vaccination or scheduled within 14 days after other vaccination (e.g., measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever; influenza vaccine in nasal form)
* Investigational research agents within 30 days prior to first study vaccination
* Any vaccines that are not live attenuated vaccines within 14 days prior to first study vaccination
* Allergy treatment with antigen injections within 30 days prior to first vaccination or scheduled within 14 days after vaccination
* Received investigational research agents within 30 days prior to first vaccination
* Current tuberculosis (TB) prophylaxis or therapy
* Recreational cocaine or methamphetamine use within the last 12 months prior to first study vaccination
* Clinically significant medical condition, abnormal physical exam findings, abnormal laboratory results, or past medical history that may affect current health. More information about this criterion can be found in the protocol.
* Any medical, psychiatric, social, or job-related condition that would interfere with the study
* Serious adverse reaction to vaccines. Participants who have had an adverse reaction to pertussis vaccine as a child are not excluded.
* Hypersensitivity to eggs or egg products
* Electrocardiogram (ECG) with clinically significant findings. More information about this criterion can be found in the protocol.
* Risk factors for heart disease. More information about this criterion can be found in the protocol.
* History of or current heart disease. More information about this criterion can be found in the protocol.
* Autoimmune disease or immunodeficiency
* Active syphilis infection. Participants with fully treated syphilis at least 6 months prior to study entry are not excluded.
* Unstable asthma. More information about this criterion can be found in the protocol.
* Diabetes mellitus type 1 or 2. Participants with a history of isolated gestational diabetes are not excluded.
* History of thyroid removal or of thyroid disease requiring treatment in the 12 months prior to study entry
* Serious angioedema within the past 3 years or requiring medication within 2 years of study entry
* Hypertension that is not well-controlled
* Body mass index (BMI) of 40 or more
* Bleeding disorder
* Cancer. Participants with surgically removed cancer that is unlikely to recur are not excluded.
* Seizure disorder requiring medication within the last 3 years
* Absence of spleen
* Certain abnormal laboratory values
* Psychiatric condition that would interfere with compliance with the protocol
* Other conditions that, in the opinion of the investigator, would interfere with the study
* Pregnancy or breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2008-11; Primary Completion 2010-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Signs and symptoms of local and systemic reactogenicity, laboratory measures of safety, and adverse events | Measured throughout study

SECONDARY OUTCOMES:
T-cell responses as detected by HIV-1 specific interferon-gamma/interleukin-2 intracellular cytokine staining | Measured 2 weeks following the fourth and fifth vaccinations
HIV-1-specific neutralizing and binding antibody assays | Measured 2 weeks following the fourth and fifth vaccinations

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Gray, Study Chair — University of the Witswatersrand; Kenneth Mayer, Study Chair — Fenway Community Health
Locations (4):
- United States (2):
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Fenway Health (FH) CRS, Boston, Massachusetts
- South Africa (2):
  - Soweto HVTN CRS, Johannesburg, Gauteng
  - Emavundleni CRS, Cape Town, Western Cape

REFERENCES:
- [Background] Hanke T, McMichael AJ, Dorrell L. Clinical experience with plasmid DNA- and modified vaccinia virus Ankara-vectored human immunodeficiency virus type 1 clade A vaccine focusing on T-cell induction. J Gen Virol. 2007 Jan;88(Pt 1):1-12. doi: 10.1099/vir.0.82493-0. PMID 17170430
- [Background] Verrier F, Burda S, Belshe R, Duliege AM, Excler JL, Klein M, Zolla-Pazner S. A human immunodeficiency virus prime-boost immunization regimen in humans induces antibodies that show interclade cross-reactivity and neutralize several X4-, R5-, and dualtropic clade B and C primary isolates. J Virol. 2000 Nov;74(21):10025-33. doi: 10.1128/jvi.74.21.10025-10033.2000. PMID 11024131
- [Background] Williamson C, Morris L, Maughan MF, Ping LH, Dryga SA, Thomas R, Reap EA, Cilliers T, van Harmelen J, Pascual A, Ramjee G, Gray G, Johnston R, Karim SA, Swanstrom R. Characterization and selection of HIV-1 subtype C isolates for use in vaccine development. AIDS Res Hum Retroviruses. 2003 Feb;19(2):133-44. doi: 10.1089/088922203762688649. PMID 12639249
- [Derived] Gray GE, Mayer KH, Elizaga ML, Bekker LG, Allen M, Morris L, Montefiori D, De Rosa SC, Sato A, Gu N, Tomaras GD, Tucker T, Barnett SW, Mkhize NN, Shen X, Downing K, Williamson C, Pensiero M, Corey L, Williamson AL. Subtype C gp140 Vaccine Boosts Immune Responses Primed by the South African AIDS Vaccine Initiative DNA-C2 and MVA-C HIV Vaccines after More than a 2-Year Gap. Clin Vaccine Immunol. 2016 Jun 6;23(6):496-506. doi: 10.1128/CVI.00717-15. Print 2016 Jun. PMID 27098021